CLINICAL TRIAL: NCT00617838
Title: Prevention of Celiac Disease in Children at Genetic Risk - Optimized Introduction of Gluten and Follow-up of Immunization
Brief Title: Celiac Disease Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other); University of Turku (Other); Finnish Institute for Health and Welfare (Other Government); Päivikki and Sakari Sohlberg Foundation, Finland (Other); Kätilöopisto Maternity Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KUH5021612
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Celiac Disease
Keywords: Celiac disease; genetic risk; gluten introduction; predicting antibodies
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Optimization of gluten introduction by nutritional councelling
  Interventions: Other: Optimal gluten introduction
- 2 (No Intervention): No specific nutritional councelling. Follow-up of gluten introduction

INTERVENTIONS:
Other: Optimal gluten introduction — Optimization of gluten introduction by nutritional counselling
  Arms: 1

SUMMARY:
Celiac disease is an autoimmune disease induced by wheat gluten. Destruction of epithelial cells and microvilli on gut mucosa is causing a "flat mucosa" and an absorption defect. The diagnosis is based on typical microscopical finding in biopsy specimens but serum antibodies to tissue transglutaminase and certain gliadin peptides are strongly associated with the pathology. Severe diarrhoea associated with growth disturbance in infancy was historically characterising the disease but is nowadays rare. Clinically more mild forms including silent disease are very common. Studies based on antibody screening and biopsies done in autoantibody positive subjects have confirmed a frequency of about 1-2% in adult population. Undiagnosed disease is associated with deficiencies of nutrients and vitamins leading to various chronic symptoms like anaemia, osteoporosis and general fatigue. It has also been recently found that undiagnosed celiac disease may be associated with general underachievement in society probably associated with common psychological symptoms like fatigue and depression during the adolescence. The disease is treated by complete elimination of wheat, rye and barley in the diet, which is laborious and causing considerable extra costs in nutrition.

Much progress has been recently made in understanding of the genetic background and immune markers associated with the disease as well as in understanding those patterns of gluten introduction in infancy, which might be connected to a high disease risk. Our aim in this study is in the first phase to identify children at high genetic risk (around 10%) and in a follow-up study to define:

1. Are the age, dose of gluten and presence of simultaneous breast feeding at the introduction of gluten associated with the risk of celiac disease?
2. Is it possible to decrease the frequency of celiac disease by nutritional counselling?
3. Is it possible to predict development of celiac disease by immunological tests before the development of mucosal lesion

If we can confirm, that optimising the conditions at the introduction of wheat gluten in infancy diet significantly reduces the disease incidence, will this have an important effect on the nutritional recommendations concerning the diet in infancy. Combining genetic screening and immunological tests might also offer a way to reduce the frequency of celiac disease and help in early diagnosis and organisation of an adequate treatment

ELIGIBILITY:
Inclusion Criteria:

* Presence of HLA-risk alleles DQA1*05 and DQB1*02

Exclusion Criteria:

* Lack of these HLA risk alleles

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2007-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
development of transglutaminase antibodies | 2-4 year age

SECONDARY OUTCOMES:
gliadin peptide antibodies | 2-4 years
mucosal biopsy in TGA positive childre | 2-4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jorma Ilonen, MD, Principal Investigator — University of Eastern Finland
Locations (1):
- Kuopio University Hospital, Kuopio, Finland